CLINICAL TRIAL: NCT02173366
Title: Preliminary Investigation of Civic Engagement as a Novel Approach to Behavior Change and Body Weight Improvement in African American Females
Brief Title: Change Clubs for African American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Boston Nutrition Obesity Research Center (administered by Boston Medical Center) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Prevention
Other Study IDs: 11244
Record Dates: First submitted 2014-06-10; First posted 2014-06-25 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Obesity; Cardiovascular Disease
MeSH Terms: conditions — Obesity; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Change Club Intervention (Experimental)
  Interventions: Behavioral: Change Club Intervention

INTERVENTIONS:
Behavioral: Change Club Intervention

SUMMARY:
African American women have among the highest rates of overweight and obesity and few meet dietary or physical activity guidelines. The investigators seek to develop a new intervention strategy that will help alleviate health disparities, thereby improving quality of life, health care costs, and disease burden. The African American Collaborative Obesity Research Network (AACORN) recommends an eco-social, community-engaged approach to behavior change that is in line with cultural values of interconnectedness and care for others. The purpose of this study is to operationalize the AACORN paradigm to promote improvements in weight status and health through a civic engagement approach. To achieve this, participants will meet in church-based Change Clubs and be led through a 6 month curriculum, which includes both lessons in cardiovascular risk reduction and a civic engagement project. Civic engagement may lead to change in individual health behaviors by increasing self-regulation and self-efficacy. The investigators will measure club members' adherence to the Change Club intervention, defined as average number of sessions attended, retention in the clubs, satisfaction with the Change Club experience and achievement of at least 50% of self-identified benchmarks for community change within 6 months. In addition the investigators will compare anthropometric factors, diet and physical activity behaviors, blood pressure, cardiorespiratory fitness, and psychosocial factors before and after participation in the Change Club intervention.

ELIGIBILITY:
Inclusion Criteria:

* female;
* age 30-70 years;
* self-identified as African American;
* English-speaking;
* BMI ≥25.0;
* currently sedentary (not meeting Physical Activity Guidelines for Americans);
* safe to initiate moderate physical activity per the PAR-Q.

Exclusion Criteria:

* failure to provide informed consent;
* participation in any other lifestyle modification program;
* current use of either prescription or over-the-counter weight loss medications;
* inability to communicate due to severe,
* uncorrectable hearing loss or speech disorder;
* severe visual impairment (if it precludes completion of assessments and/or intervention);
* planning to move outside of area within 6 months;
* pregnancy (since weight loss, the primary outcome, is inadvisable in this population).

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-12; Primary Completion 2015-11 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Weight from Pre to Post-Intervention (6 Months) | pre-post; participants will be followed for the 6-month intervention period
  Body weight will be measured in triplicate to the nearest 0.5 kg using a digital floor scale (Seca 876).

SECONDARY OUTCOMES:
Change in Diet from Pre to Post-Intervention (6 Months) | pre-post; participants will be followed for the 6-month intervention period
  Two 24-hour recalls (1 weekday and 1 weekend day) will be collected. Data will be entered into the Nutrition Data System for Research (NDSR). Nutrient and food group calculations will be performed using the NDSR software.
Change in Physical Activity Level from Pre to Post-Intervention (6 Months) | pre-post; participants will be followed for the 6-month intervention period
  Physical activity levels will be measured objectively using accelerometers (ActiGraph GT3X worn for 7 days) and by self-report (7-Day Physical Activity Recall).
Change in Blood Pressure from Pre to Post-Intervention (6 Months) | pre-post; participants will be followed for the 6-month intervention period
  Blood pressure will be measured to the nearest 1mm Hg using a validated automated monitor (Omron HEM-705CP), using American Heart Association guidelines.
Change in Cardiorespiratory Fitness Level from Pre to Post-Intervention (6 Months) | pre-post; participants will be followed for the 6-month intervention period
  Cardiovascular fitness will be measured using the Rockport 1-mile walk test. Participants will walk a flat, 1-mile course as fast as possible without running. Heart rate will be measured immediately after. VO2max will be estimated from validated formulas using 1-mile walk time, gender, age, body weight, and ending heart rate.
Change in Self-Efficacy from Pre to Post-Intervention (6 Months) | pre-post; participants will be followed for the 6-month intervention period
  Self-efficacy will be assessed the Weight Efficacy Life-Style Questionnaire (Clark 1991). The exercise self-efficacy scale contains 5 items measuring confidence in ability to exercise under various challenges.
Change in Collective Efficacy from Pre to Post-Intervention (6 Months) | pre-post; participants will be followed for the 6-month intervention period
  Collective efficacy will be measured using an adapted 8-item Likert style scale (Sampson, Raudebush, & Earls 1997) that examines the extent to which individuals in a neighborhood or community trust and help others.
Change in Percent Body Fat from Pre to Post-Intervention (6 Months) | pre-post; participants will be followed for the 6-month intervention period
  Percent body fat will be measured by bioelectric impedance using a Tanita TBF-410 Bioelectric Impedance Body Composition Analyzer.
Change in Perceived Stress from Pre to Post-Intervention (6 Months) | pre-post; participants will be followed for the 6-month intervention period
  Perceived stress will be measured using the validated 14-item Perceived Stress Scale (Cohen 1983).
Change in Level of Civic Engagement from Pre to Post-Intervention (6 Months) | pre-post; participants will be followed for the 6-month intervention period
  We will use the Civic Engagement Scale (Doolittle and Faul 2013) to assess civic engagement.
Change in Level of Self-Regulation from Pre to Post-Intervention (6 Months) | pre-post; participants will be followed for the 6-month intervention period
  Self-regulation will be measured using a scale developed by Saelens et al. (2000) to measure self-regulatory skill usage for exercise and for controlled eating.

OTHER OUTCOMES:
Adherence | attendance will be monitored throughout the 6-month intervention period
Retention | participant retention will be monitored throughout the 6-month intervention period

CONTACTS AND LOCATIONS:
Locations (1):
- Friedman School of Nutrition, Tufts University, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Brown AG, Hudson LB, Chui K, Metayer N, Lebron-Torres N, Seguin RA, Folta SC. Improving heart health among Black/African American women using civic engagement: a pilot study. BMC Public Health. 2017 Jan 24;17(1):112. doi: 10.1186/s12889-016-3964-2. PMID 28118823